CLINICAL TRIAL: NCT00330317
Title: Neoadjuvant Hormone Therapy for Postmenopausal Women With HR+ Primary Breast Cancer: A Multi-center Study to Determine the Optimum Length of Treatment With Letrozole on Tumour Regression to Permit Breast Conserving Surgery.
Brief Title: Safety and Efficacy of Hormone Therapy With Letrozole in Postmenopausal Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345EGB07
Record Dates: First submitted 2006-05-24; First posted 2006-05-26 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: Letrozole; Breast Conserving Surgery; NeoAdjuvant; Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Letrozole (Experimental)
  Interventions: Drug: letrozole

INTERVENTIONS:
Drug: letrozole — 2.5mg letrozole once-daily
  Other Names: Femara, FEM345

SUMMARY:
The aim of this study is to assess the safety and efficacy of neoadjuvant hormone therapy with letrozole in postmenopausal women with estrogen- and/or progesterone-receptor positive primary breast cancer on tumour regression to permit breast conserving surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women able to comply with the protocol requirements with confirmed primary invasive breast cancer whose tumours are estrogen-and/or progesterone-receptor positive
2. Clinical stage T2 or >T2 tumours which in the investigators' opinion would not be eligible for breast-conserving surgery. The nodal status will be evaluated by palpation and/or ultrasound.
3. Postmenopausal status defined by one of the following:

   * Women with an intact uterus AND

     * ≥ 55 years of age, OR
     * < 55 years of age without menses for the last 5 years, OR
     * < 55 years of age and have not had menses for at least the last 12 months (but have had menses in the last 5 years) and have postmenopausal levels of follicle-stimulating hormone.
   * Women without an intact uterus AND

     * ≥ 55 years of age, OR
     * < 55 years of age and postmenopausal levels of follicle-stimulating hormone
   * Both ovaries removed (prior to the diagnosis of breast cancer).
4. Tumour measurable by clinical examination, mammography and ultrasound
5. Adequate bone marrow function as shown by:

   * WBC ≥ 3.5 x 10^9/L
   * ANC ≥ 1.5 x 10^9/L
   * Platelets ≥ LLN
   * Hb > 10 g/dL

Exclusion Criteria:

1. Multifocal disease (cancer that starts in several different sites)
2. Patients with bilateral breast tumours.
3. Patients who are eligible for breast conserving surgery.
4. Evidence of inflammatory breast cancer or distant metastasis.
5. Simultaneous anti-cancer treatments such as chemotherapy, immunotherapy/biological response modifiers, endocrine therapy (including steroids), bisphosphonate therapy and radiotherapy. NOTE: Bisphosphonate therapy for osteoporosis is NOT excluded, and can be continued. Patients who have received hormone replacement therapy will NOT be excluded if it is discontinued at least 2 weeks before starting the study.

The following additional treatments are NOT allowed during the treatment phase of the study:

* Any other anti-cancer therapy
* Hormone replacement therapy.
* Estrogen cream (including any intra-vaginal preparation).
* Steroids other than creams or inhalers.
* Megestrol acetate for the treatment of hot flushes.
* Radiation therapy.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2006-02; Primary Completion 2010-03 (Actual); Study Completion 2010-11-16 (Actual)

PRIMARY OUTCOMES:
Optimum length of treatment with letrozole (2.5 mg daily) preoperatively, on tumour measured by clinical examination and breast ultrasound | 12 months

SECONDARY OUTCOMES:
Reduction in tumour volume every 2 months throughout the study | 12 months
Response rate in line with the Response Evaluation Criteria in Solid Tumors criteria | 12 months
Long term (5-year) local recurrence rate | 5 years
Safety and tolerability of the treatment prior to surgery | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (20):
- United Kingdom (20):
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, Brighton
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Crewe
  - Novartis Investigative Site, Dundee
  - Novartis Investigative Site, East Sussex
  - Novartis Investigative Site, Epping
  - Novartis Investigative Site, Farnworth
  - Novartis Investigative Site, Gateshead
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Hants
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Luton
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Newcastle
  - Novartis Investigative Site, Poole
  - Novartis Investigative Site, Saint Leonards-on-Sea
  - Novartis Investigative Site, West Smithfield

REFERENCES:
- [Result] Carpenter R, Doughty JC, Cordiner C, Moss N, Gandhi A, Wilson C, Andrews C, Ellis G, Gui G, Skene AI. Optimum duration of neoadjuvant letrozole to permit breast conserving surgery. Breast Cancer Res Treat. 2014 Apr;144(3):569-76. doi: 10.1007/s10549-014-2835-8. Epub 2014 Feb 23. PMID 24562823